CLINICAL TRIAL: NCT04305860
Title: Acceptance of Different Types of Thickeners, With and Without Flavoring, in Patients With Dysphagia
Brief Title: Acceptance of Different Thickeners in Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Principal Investigator, Alfonso Vidal Casariego, Principal Investigator, Complexo Hospitalario Universitario de A Coruña
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-527
Record Dates: First submitted 2020-03-03; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Dysphagia; Dysphagia, Oropharyngeal
Keywords: Thickener; Flavoring; Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Flavoring Agents; xanthan gum

STUDY DESIGN:
Intervention Model Description: Pilot study of nutritional intervention, randomized, and controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Modified starch without flavoring (Active Comparator): Patients thicken water with modified starch during 3 days of hospitalization. They evaluate the organoleptic characteristics of the thickened liquid and register the volume of water intake.
  Interventions: Dietary Supplement: Modified starch without flavoring
- Modified starch with flavoring (Active Comparator): Patients thicken water with modified starch adding any of 5 kinds of flavorings "Bi1 aromas" during 3 days of hospitalization. They evaluate the organoleptic characteristics of the thickened liquid and register the volume of water intake.
  Interventions: Dietary Supplement: Mofidied starch with Bi1 aromas
- Xanthan gum without flavoring (Active Comparator): Patients thicken water with xanthan gum during 3 days of hospitalization. They evaluate the organoleptic characteristics of the thickened liquid and register the volume of water intake.
  Interventions: Dietary Supplement: Xanthan gum without flavoring
- Xanthan gum with flavoring (Active Comparator): Patients thicken water with xanthan gum adding any of 5 kinds of flavorings "Bi1 aromas" during 3 days of hospitalization.They evaluate the organoleptic characteristics of the thickened liquid and register the volume of water intake.
  Interventions: Dietary Supplement: Xanthan gum with Bi1 aromas

INTERVENTIONS:
Dietary Supplement: Modified starch without flavoring — Each patient of this group receives the thickener during three days of hospitalization
  Arms: Modified starch without flavoring
Dietary Supplement: Mofidied starch with Bi1 aromas — Each patient of this group receives the thickener and 5 flavorings during three days of hospitalization
  Arms: Modified starch with flavoring
Dietary Supplement: Xanthan gum without flavoring — Each patient of this group receives the thickener during three days of hospitalization
  Arms: Xanthan gum without flavoring
Dietary Supplement: Xanthan gum with Bi1 aromas — Each patient of this group receives the thickener and 5 flavorings during three days of hospitalization
  Arms: Xanthan gum with flavoring

SUMMARY:
Randomized, controlled, pilot study of nutritional intervention to evaluate the acceptance to different kinds of thickeners, with and without the addition of flavoring.

DETAILED DESCRIPTION:
Background:

In patients with dyaphagia the modification of viscosity of oral liquids with thickeners ia needed to guarantee an effective and safe swallowing, and to ensure a proper state of hydration. There are two types of thickeners: thickeners obtained from modified starch or from food gums (suchxanthan gum)

Aim:

To evaluate the acceptance of different types of thickeners, with and without the addition of flavorings, and their relationship with water intake.

Methods:

Randomized, controlled, pilot study of nutritional intervention. Forty hospitalized patients with oropharyngeal dysphagia were randomized to 4 parallel groups: modified starch without flavoring, modified starch with flavoring, xanthan gum without flavoring, xanthan gum with flavoring. Each patient was asked to assess the odor, taste, appearance, and overall valoration of the thickened liquid with the different preparations, using a structured questionnaire. The number of glasses consumed by the patient over 3 consecutive days was also recorded to calculate de volume of liquid they consumed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oropharyngeal dysphagia for liquids diagnosed before admission or during hospitalization and who need thickener.

Exclusion Criteria:

* Patients with expected hospital length of stay less than 24 hours.
* Patients with food allergy to any of the ingredients of the thickener or flavorings used in the study.
* Patients with cognitive impairment that prevents collaborating in obtaining data.
* Patients in terminal situations, in which death is expected in the following hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Hydratation | 3 days during hospitalization
  Volume of water ingested (ml)
Taste | 3 days during hospitalization
  Semiquantitative scale of Punctuation of taste: 1-5 points (1: very bad; 2: bad; 3: intermediate; 4: Good; 5: very good).
Odor | 3 days during hospitalization
  Semiquantitative scale of Punctuation of odor: 1-5 points (1: very bad; 2: bad; 3: intermediate; 4: Good; 5: very good).
Appearance | 3 days during hospitalization
  Semiquantitative scale of Punctuation of appearance: 1-5 points (1: very bad; 2: bad; 3: intermediate; 4: Good; 5: very good).
Overall valoration | 3 days during hospitalization
  Quantiative scale of Punctuation: 0-10 points (very bad to very good).

CONTACTS AND LOCATIONS:
Locations (1):
- Alfonso Vidal-Casariego, A Coruña, La Coruna, Spain